CLINICAL TRIAL: NCT04702711
Title: Experiences of Anger in Patients in Primary Health Care With Symptoms of Generalized Anxiety - a Qualitative Study From the Perspective of Patients and Health Care Professionals
Brief Title: Experiences of Anger in Patients in Primary Health Care With Symptoms of Generalized Anxiety
Status: Recruiting | Type: Observational
Sponsor: Kronoberg County Council (Other Government)
Collaborators: Linnaeus University (Other)
Responsible Party: Sponsor
Other Study IDs: 20RGK1676
Record Dates: First submitted 2020-12-10; First posted 2021-01-11 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Generalized Anxiety; Anger; Primary Health Care
Keywords: Generalized Anxiety; Worry; Anger; Primary Health Care
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with symptoms of generalized anxiety in primary health care: Patients (18 years or older) with symptoms of generalized anxiety at a primary health care center.
  Interventions: Other: No intervention
- Health care professionals: Health care professionals working with patients with symptoms of generalized anxiety in a primary health care center.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Symptoms of generalized anxiety is common in the general population and is often treated in primary health care. Anger is an emotion that can lead to interpersonal problems but can also be an agent for justice and change. Previous research has shown a link between generalized anxiety and anger but there is a lack of qualitative research investigating how individuals with symptoms of generalized anxiety experience anger.

The aim of this research study is to increase knowledge about how anger is experienced in adult patients in primary health care with symptoms of generalized anxiety and about the experiences of health care professionals working with patients with symptoms of generalized anxiety.

DETAILED DESCRIPTION:
Symptoms of generalized anxiety is common in the general population and is often treated in primary health care. The core of the diagnostic criteria for generalized anxiety disorder (GAD) is excessive long-term worry that is difficult to control and concerns a number of events or activities. In this study we use the term "symptoms of generalized anxiety" by which we refer to these symptoms, regardless of whether the patient has a clinically established diagnosis of GAD or not.

Anger is an emotion that can lead to interpersonal problems but can also be an agent for justice and change. Previous research has shown a link between generalized anxiety and anger but there is a lack of qualitative research on how individuals with symptoms of generalized anxiety experience anger.

The aim of this research study is to increase knowledge about how anger is experienced in adult patients in primary health care with symptoms of generalized anxiety and about the experiences of health care professionals working with patients with symptoms of generalized anxiety.

The study has the following research questions:

1. How do adult patients in primary health care with symptoms of generalized anxiety experience their own anger?
2. How do health care professionals experience anger in patients in primary health care with symptoms of generalized anxiety?
3. How do health care professionals experience attitudes towards and treatment of adult patients with symptoms of generalized anxiety in primary health care with special focus on the patients' anger?

Patients with symptoms of generalized anxiety and health care professionals at primary health care centers are interviewed (se section on eligibility). The goal is to include 15-20 patients and 15-20 health care professionals. A questionnaire with background questions is completed and the interviews follow an interview guide. The background questionnaire and interview guide differ between patients and health care professionals. The interviews are audio recorded and transcribed into text. The data is analyzed using thematic analysis according to the guidelines given by Braun and Clarke (2006; 2013).

ELIGIBILITY:
Patients with symptoms of generalized anxiety

Inclusion Criteria:

* Clinically significant level of symptoms of generalized anxiety which is confirmed by a self-rated diagnose of GAD on the questionnaire GAD-Q-IV (Newman et al., 2002; Moore et al., 2014). The questions of the GAD-Q-IV correspond to the A, B, C and D criteria of GAD in Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
* Sufficient knowledge in Swedish to be able to answer questionnaires and take part in an interview.
* If the patient receives any medical or psychological treatment for generalized anxiety this should be recently started and/or not yet have led to any notable decrease of symptoms. In the case of pharmacological treatment this should not be associated with more extensive psychological side-effects.

Exclusion Criteria:

* Severe psychiatric difficulties where the patient needs specialized psychiatric care
* Known brain-injury or symptoms of dementia
* The patient is in an acute crisis
* Obvious alcohol or substance abuse

Health care professionals

Inclusion Criteria:

* Have a health care profession and work at a primary health care center.
* Current working experience of at least one year at a primary health care center which included contact with patients with symptoms of generalized anxiety

Exclusion Criteria:

- Being at the primary health care center in the role of an external student

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study has two populations:
  * Patients with symptoms of generalized anxiety in primary health care.
  * Health care professionals working in primary health care who come into contact with or treat patients with symptoms of generalized anxiety
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patients' experiences of anger | Up to 6 months after enrollment
  Qualitative interview with adult patients with symptoms of generalized anxiety
Health care professionals' experiences of anger in adult patients with symptoms of generalized anxiety | Up to 6 months after enrollment
  Qualitative interview with health care professionals
Health care professionals' experiences of attitudes towards and treatment of adult patients with symptoms of generalized anxiety | Up to 6 months after enrollment
  Qualitative interview with health care professionals

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Carlsson, Phd, Study Director — Regional Department of Competence in Family Medicine and Primary Health Care, Region Kronoberg
Locations (1):
- Region Kronoberg, Vaxjo, Sweden

IPD SHARING:
Plan to Share IPD: No